CLINICAL TRIAL: NCT04822467
Title: SQ53 Disinfectant Wipes for Prevention of Catheter Related Blood Stream Infection in Patients Receiving Home Parenteral Nutrition: A Single Blind Randomized Placebo-controlled Clinical Trial
Brief Title: SQ53 Disinfectant Wipes for Prevention of CRBSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: JVS Products, Ltd. (Unknown)
Responsible Party: Principal Investigator, Donald Kirby, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CC-SQ53
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Catheter-related Bloodstream Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard Wipe (Active Comparator): Participants will receive a supply of ethanol-based wipes for daily use
  Interventions: Device: Ethanol Wipe
- SQ53 Wipe (Experimental): Participants will receive a supply of SQ53 wipes for daily use.
  Interventions: Device: SQ53 Wipe

INTERVENTIONS:
Device: SQ53 Wipe — SQ53-based wipe to be used by the participant daily or upon dressing change
  Arms: SQ53 Wipe
Device: Ethanol Wipe — Ethanol-based wipe to be used by the participant daily or upon dressing change
  Arms: Standard Wipe

SUMMARY:
SQ53 is a novel antimicrobial, sporicidal solution that is based on a platform of quaternary ammonium chloride compounds. It has been tested against a wide range of bacteria, viruses, spores and fungal pathogens. Extensive laboratory testing has demonstrated the effectiveness of SQ53 impregnated wipes in cleaning surfaces including catheters over a 24 hour plus time period. SQ53 also received an in vitro evaluation of the irritancy potential using a tissue engineered human skin model and was found to have no potential for skin irritation. SQ53 is available as a sterilized pack with a single wipe inside. The pack is easy to open by tearing off the top end and presenting the contents to the operator to remove under sterile conditions.

The current study will be a randomized single-blinded placebo-controlled clinical trial for SQ53 wipes intended for catheter cleaning in patients receiving home parenteral nutrition.

DETAILED DESCRIPTION:
Parenteral nutrition (PN) therapy is an essential component of medical management of patients suffering from intestinal failure. Depending on the underlying etiology and the type of intestinal failure, the duration of parenteral nutrition therapy could range from several weeks to several years, although a substantial proportion of these patients also require lifelong parenteral nutrition support. These patients continue the infusion of PN at their homes and are managed by the Cleveland Clinic's Home PN support team. These patients require Central Venous Catheters (CVC) for prolonged period of time for infusion of parenteral nutrition. The two most commonly used central catheters for TPN infusion are the Peripherally Inserted Central Catheter (PICC) and Tunneled CVCs. Catheter related blood stream infection (CRBSI) is a major complication of long-term CVCs. CRBSI is associated with high morbidity, mortality and healthcare cost. Additionally, CRBSI can also lead to an interruption in nutrient delivery, loss of work and productivity, premature vascular access device removal, and poor quality of life.

Prevention of CRBSI is an important component of clinical management of patients receiving home PN therapy. Several strategies have been adopted to reduce the incidence of CRBSI. A heparin lock solution was used in the past for many years; however, current nutrition society guidelines recommend normal saline locks instead of heparin locks. Published data has suggested that heparin locks have not proven to have a substantial effect on CRBSI prevention, and it paradoxically increases the infection risk due to biofilm production. Antibiotic locks have also been used, although this practice is largely not preferred due to increased risk of infections with resistant microorganisms. Taurolidine is another lock solution which has been studied in the countries outside the United States such as Canada; however, it has not been approved for the use in the U.S. yet.1

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring home parenteral nutrition support via PICC line or tunneled CVC.

Exclusion Criteria:

* Age less than 18 years
* Women known to be pregnant
* Women of childbearing age who are planning a pregnancy
* Women who are breastfeeding
* Patients who will not be managed by Cleveland Clinic HPN service
* Patients who refuse to use disinfectant wipes daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Kirby, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Wipe | SQ53 Wipe
Started | 29 | 30
Completed | 29 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Wipe | SQ53 Wipe | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.7 (15) | 51.7 (17.6) | 52.2 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 47
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27 | 28 | 55
  African American | 1 | 2 | 3
  Asian or Pacific Islander | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Catheter-Related Blood Stream Infections (CRBSI) at 6 Months
Description: Reduction in the number of CRBSI experienced by participants over a six month period (1000 days)
Time Frame: 6 months
Population: Data analysis was done on all subjects enrolled as well as those that met the protocol defined compliance rates.
  Subjects were removed due inability to continue with the protocol (moving to different Home Parenteral Nutrition service or not following treatment guidelines)
Measure: Mean (Inter-Quartile Range); unit: Infections per 1000 days with catheter
Arm/Group | Standard Wipe | SQ53 Wipe
Number analyzed (Participants) | 29 | 30
Infections per 1000 days with catheter
  Intention to Treat | 1.98 [1.17 to 3.34] | 2.09 [1.21 to 3.59]
  Met Protocol Compliance Definitions: number analyzed (Participants) | 26 | 24
  Met Protocol Compliance Definitions | 1.73 [0.96 to 3.13] | 1.02 [0.46 to 2.28]

2. Secondary Outcome: Catheter Exchange Rates
Description: Reduction in catheter exchange rates by participants over 1000 days
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: Exchanges per 1000 days with Catheter
Arm/Group | Standard Wipe | SQ53 Wipe
Number analyzed (Participants) | 29 | 30
Exchanges per 1000 days with Catheter
  Intention to Treat | 1.41 [0.76 to 2.62] | 1.61 [0.86 to 2.98]
  Met Protocol Compliance Definitions: number analyzed (Participants) | 26 | 24
  Met Protocol Compliance Definitions | 1.26 [0.63 to 2.52] | 0.68 [0.26 to 1.82]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subject reported events
Arm/Group | Standard Wipe | SQ53 Wipe
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 1/29 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Wipe (N=29) | SQ53 Wipe (N=30)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT04822467/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/67/NCT04822467/ICF_001.pdf